CLINICAL TRIAL: NCT05308680
Title: A Prospective Study for Myocardial Injury After BNT162b2 mRNA COVID-19 Fourth Dose Vaccination Among Israeli Health Care Workers
Brief Title: Myocardial Injury After BNT162b2 mRNA COVID-19 Fourth Dose Vaccination Among Israeli Health Care Workers
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Tal Hasin, Head of Heart Failure Unit, Jesselson Integrated Heart Center,, Shaare Zedek Medical Center
Other Study IDs: 001
Record Dates: First submitted 2022-03-31; First posted 2022-04-04 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Myocardial Injury; Vaccine Adverse Reaction; COVID-19
Keywords: myocardial injury; vaccine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: BNT162b2 — Administration of the fourth dose BNT162b2 mRNA vaccine (Pfizer-BioNTech) against COVID-19

SUMMARY:
The aim of the study is to prospectively evaluate the incidence of myocardial injury after the administration of the fourth dose BNT162b2 mRNA vaccine (Pfizer-BioNTech) against COVID-19.

DETAILED DESCRIPTION:
Population-based retrospective studies suggest an association between BNT162b2 (Pfizer-BioNTech) vaccination against coronavirus disease 2019 (COVID-19) and myocarditis. While the overall incidence of myocarditis is estimated to be 2.13 per 100,000 persons, the incidence of myocardial injury and subclinical myocarditis may be higher. Adult health care workers who received the BNT162b2 vaccine in two Israeli hospitals (SZMC and Shamir) during the fourth dose campaign had blood samples taken for high-sensitivity cardiac troponin (hs-cTn) measurement at the time of vaccine administration and after 2-4 days. Post-vaccine myocardial injury was defined as hs-cTn elevation above the 99th percentile upper reference limit and >50% increase from the first measurement. Participants with evidence of myocardial injury underwent assessment for possible myocarditis including electrocardiogram and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult health care workers (≥18 years old)

Exclusion Criteria:

* Acute coronary syndrome, peri/myocarditis, cardiac catheterization, cardiac surgery, cardiac ablation, or any other invasive cardiac procedure within 14 days prior to study enrollment.
* Chronic renal failure (creatinine clearance ≤30 mL/min), or dilated or hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult health care workers who received the BNT162b2 vaccine (Pfizer-BioNTech) during the fourth dose campaign
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Myocardial Injury | 2-4 days after vaccine administration
  Myocardial injury was defined as high sensitivity cardiac troponin elevation above the 99th percentile upper reference limit and >50% increase from baseline measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare zedek MC, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levi N, Moravsky G, Weitsman T, Amsalem I, Bar-Sheshet Itach S, Algur N, Lapidus I, Mitz O, Glikson M, Wiener-Well Y, Hasin T. A prospective study on myocardial injury after BNT162b2 mRNA COVID-19 fourth dose vaccination in healthy persons. Eur J Heart Fail. 2023 Feb;25(2):313-318. doi: 10.1002/ejhf.2687. Epub 2022 Sep 28. PMID 36097844